CLINICAL TRIAL: NCT03764813
Title: Fetal Hemoglobin Levels and Umbilical Cord or Adult Blood RBC Transfusions in Preterm Neonates.
Brief Title: Cord Blood Transfusion In Preterm Neonates (CB-TrIP)
Acronym: CB-TrIP
Status: Completed | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TEOFILI LUCIANA, Medical Director of the UNICATT Cord Blood Bank, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 22139/18ID:1916
Record Dates: First submitted 2018-11-22; First posted 2018-12-05 (Actual); Results first posted 2020-04-24 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-08

CONDITIONS: Premature Infant Disease; Transfusion Related Complication; Fetal Hemoglobin
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 80-100 microL of capillary blood for HbF assessment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Repeated transfusions have been associated with very poor outcome of preterm infants. Fetal hemoglobin (HbF) and adult Hb (HbA) have different affinity for oxygen. The high level of adult Hb may contribute to exacerbating the oxidative damage responsible for prematurity diseases. The investigators hypothesized that transfusing red blood cells (RBC) obtained from allogeneic cord blood (CB) of healthy full-term babies (which contains almost exclusively HbF) may prevent the non-physiological decrease of HbF in premature neonates, likewise protecting them from oxygen radical diseases. Cord blood transfusion in preterms - CB TRIP - is a monocentric prospective nonrandomized study aimed to monitor HbF levels in preterm neonates receiving RBC transfusions from either umbilical blood of full-term healthy babies (CB-RBC) and/or from adult donors (A-RBC).

DETAILED DESCRIPTION:
Preterm neonates enrolled in this study are monitored for the level of HbF on capillary blood samples, from birth to the week 32 of postmenstrual age (PMA). To fulfill the RBC transfusion requirements, RBC concentrates obtained from umbilical blood of full-term healthy babies are utilized, if available; otherwise, RBC concentrates from adult donors are assigned. For every week of PMA, neonates undergo a minimum of three HbF determinations, and the median values are considered.

ELIGIBILITY:
Inclusion Criteria:

preterm neonates born at PMA ≤30 weeks and/or with birth weight ≤1000 g born at the delivery room of Fondazione Policlinico Universitario A. Gemelli candidate to receive one or more RBC unit transfusion.

Exclusion Criteria:

One or more of the following criteria Maternal-fetal immunization Hydrops fetalis Major congenital malformations associated or not with genetic syndromes Previous transfusions Hemorrhage at birth Congenital infections (such as infections from TORCH complex) Out-born infants The health care team deems it inappropriate to approach the infant's family for informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The CB TRIP trial enrolls preterm neonates born before the 30th week of gestation and/or neonates with birth weight <1000 grams, admitted to the NICU of Policlinico Gemelli, and candidate to receive one or more RBC transfusions. These characteristics (birth <28 weeks of gestation and birth weight <1000 grams) identify a very fragile population, with significant early mortality and morbidity and high risk for lifelong invalidating consequences.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2019-08-02 (Actual); Study Completion 2019-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Teofili, MD, PhD, Principal Investigator — Fondazione Policlinico Agostino Gemelli IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM
  - Fondazione Policlinico Universitario A.Gemelli IRCCS, Rome

REFERENCES:
- [Background] Bianchi M, Papacci P, Valentini CG, Barbagallo O, Vento G, Teofili L. Umbilical cord blood as a source for red-blood-cell transfusion in neonatology: a systematic review. Vox Sang. 2018 Nov;113(8):713-725. doi: 10.1111/vox.12720. Epub 2018 Oct 16. PMID 30328121
- [Background] Bianchi M, Giannantonio C, Spartano S, Fioretti M, Landini A, Molisso A, Tesfagabir GM, Tornesello A, Barbagallo O, Valentini CG, Vento G, Zini G, Romagnoli C, Papacci P, Teofili L. Allogeneic umbilical cord blood red cell concentrates: an innovative blood product for transfusion therapy of preterm infants. Neonatology. 2015;107(2):81-6. doi: 10.1159/000368296. Epub 2014 Nov 15. PMID 25401961
- [Background] Stutchfield CJ, Jain A, Odd D, Williams C, Markham R. Foetal haemoglobin, blood transfusion, and retinopathy of prematurity in very preterm infants: a pilot prospective cohort study. Eye (Lond). 2017 Oct;31(10):1451-1455. doi: 10.1038/eye.2017.76. Epub 2017 May 26. PMID 28548651
- [Background] dos Santos AM, Guinsburg R, de Almeida MF, Procianoy RS, Leone CR, Marba ST, Rugolo LM, Fiori HH, Lopes JM, Martinez FE; Brazilian Network on Neonatal Research. Red blood cell transfusions are independently associated with intra-hospital mortality in very low birth weight preterm infants. J Pediatr. 2011 Sep;159(3):371-376.e1-3. doi: 10.1016/j.jpeds.2011.02.040. Epub 2011 Apr 13. PMID 21489555
- [Background] Valieva OA, Strandjord TP, Mayock DE, Juul SE. Effects of transfusions in extremely low birth weight infants: a retrospective study. J Pediatr. 2009 Sep;155(3):331-37.e1. doi: 10.1016/j.jpeds.2009.02.026. PMID 19732577
- [Derived] Teofili L, Papacci P, Orlando N, Bianchi M, Molisso A, Purcaro V, Valentini CG, Giannantonio C, Serrao F, Chiusolo P, Nicolotti N, Pellegrino C, Carducci B, Vento G, De Stefano V. Allogeneic cord blood transfusions prevent fetal haemoglobin depletion in preterm neonates. Results of the CB-TrIP study. Br J Haematol. 2020 Oct;191(2):263-268. doi: 10.1111/bjh.16851. Epub 2020 Jun 8. PMID 32510635

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Parents of neonates with birth weight < 1000 gr and/or postmenstrual age < 30 weeks consecutively admitted to the intensive neonatal unit of Fondazione Poiliclinico Gemelli IRCCS were informed about the study and asked to paricipate.
Pre-assignment Details: Among 29 couples, 25 accepted to participate and overall 25 patients were enrolled.
Units Other Than Participants: HbF measures
Groups:
- Non Transfused: Patient not receiving transfusions
- Cord-RBC Transfusions: Patients receiving exclusively allogeneic top up transfusions obtained from healthy full term neonates.
- Adult-RBC Transfusion: Patients receiving exclusively standard RBC transfusions from adult donors
- Cord- and Adult-RBC Transfusions: Patients receiving both types of transfusions
Period: From Enrollment to the Age of 32 Weeks
Arm/Group | Non Transfused | Cord-RBC Transfusions | Adult-RBC Transfusion | Cord- and Adult-RBC Transfusions
Started | 14; 127 HbF measures (Patients receiving no transfusions before the age of 32 weeks) | 3; 27 HbF measures (Patients receiving only cord-RBC transfusions before the age of 32 weeks) | 4; 38 HbF measures (Patients receiving only adult-RBC transfusions before the age of 32 weeks) | 4; 85 HbF measures (Patients receiving both adult-RBC and cord-RBCs before the age of 32 weeks)
Completed | 14; 127 HbF measures | 2; 19 HbF measures | 3; 33 HbF measures | 4; 85 HbF measures
Not Completed | 0; 0 HbF measures | 1; 8 HbF measures | 1; 5 HbF measures | 0; 0 HbF measures
Not completed — Death before the age of 32 weeks | 0 | 1 | 1 | 0
Period: From Enrollment to the Last HbF Test
Arm/Group | Non Transfused | Cord-RBC Transfusions | Adult-RBC Transfusion | Cord- and Adult-RBC Transfusions
Started | 13; 224 HbF measures (Patients receiving no transfusions before last HbF test (occurring at 36 weeks,discharge or death)) | 3; 46 HbF measures (Patients receiving only cord-RBCs before last HbF test (occurring at 36 wks,discharge or death)) | 4; 68 HbF measures (Patients receiving only adult-RBC before last HbF test (occurring at 36 wks,discharge or death)) | 5; 140 HbF measures (Patients receiving both cord and adult-RBCs before the last HbFtest(age of 36 wk,discharge or death))
Completed | 13; 224 HbF measures | 3; 46 HbF measures | 4; 68 HbF measures | 5; 140 HbF measures
Not Completed | 0; 0 HbF measures | 0; 0 HbF measures | 0; 0 HbF measures | 0; 0 HbF measures

BASELINE CHARACTERISTICS:
Population: These data refer to all patients enrolled in the study, grouped according types of transfusions received (if any) until the completion of the age of 36 weeks, discharge or death.
Units Other Than Participants: HbF measures
Groups:
- Non-Transfused: 13 patients not receiving transfusions.
- Only Cord-RBC: 3 patients receiving exclusively cord-RBC transfusions
- Only Adult-RBC: 4 patients receiving exclusively adult-RBC transfusions
- Cord- and Adult-RBC: 5 patients receiving both adult-RBC and cord-RBC transfusions
- Total: Total of all reporting groups
Arm/Group | Non-Transfused | Only Cord-RBC | Only Adult-RBC | Cord- and Adult-RBC | Total
Number analyzed (Participants) | 13 | 3 | 4 | 5 | 25
Number analyzed (HbF measures) | 224 | 46 | 68 | 140 | 478
Age, Continuous [Median (Inter-Quartile Range); unit: weeks] — Gestational age at birth (weeks)
  weeks | 30.0 [29.0 to 30.4] | 29.3 [24 to 29.3] | 28.5 [26.4 to 29.4] | 26.4 [25.2 to 28.3] | 29.4 [27.1 to 30.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 3 | 12
  Male | 8 | 1 | 2 | 2 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0 | 0 | 0
    (all) |  |  |  |  | 0
Birth weight [Median (Inter-Quartile Range); unit: grams] — Weight at birth
  grams | 1285 [1070 to 1340] | 710 [700 to 710] | 1070 [548 to 1445] | 930 [565 to 949] | 1030 [750 to 1317]
Hb at birth [Median (Inter-Quartile Range); unit: g/dL] — Hemoglobin at birth (g/dL)
  g/dL | 17.3 [14.6 to 18.0] | 16.3 [12.7 to 16.3] | 14.9 [11.9 to 16.0] | 14.2 [13.5 to 17.3] | 15.4 [13.9 to 17.5]

OUTCOME MEASURES:

1. Primary Outcome: Median Percentage of HbF at 32 Weeks of Post Menstrual Age
Description: The HbF level was determined by high-performance liquid chromatography and was expressed as percentage of total Hb, calculated as the sum of fetal and adult Hb, according to the formula: HbF= [HbF/ (FHbA1 + HbA2 + HbF)]. HbF.
Time Frame: From study entry to the completion of postmenstrual age of 32 weeks
Population: The overall amount of 264 HbF results were included in the analysis. HbF was expressed as percentage of total Hb (i.e. HbF+HbA1+HbA2)
Measure: Median (Inter-Quartile Range); unit: percentage of total Hb
Units Other Than Participants: HbF values
Groups:
- Non-transfused: 127 HbF measures obtained from 13 preterm neonates surviving until the completion of postmenstrual age of 32 weeks without receiving transfusions
- Only Cord-RBC: 19 HbF measures obtained from 2 preterm neonates surviving until the completion of postmenstrual age of 32 weeks,receiving only cord-RBC transfusions
- Only adult_RBC: 33 HbF measures obtained from 3 preterm neonates surviving until the completion of postmenstrual age of 32 weeks,receiving only adult-RBC transfusions
- Both Cord-RBC and adult_RBC: 85 HbF measures obtained from 5 preterm neonates surviving until the completion of postmenstrual age of 32 weeks,receiving both cord-RBC and adult-RBC transfusions
Arm/Group | Non-transfused | Only Cord-RBC | Only adult_RBC | Both Cord-RBC and adult_RBC
Number analyzed (Participants) | 14 | 2 | 3 | 4
Number analyzed (HbF values) | 127 | 19 | 33 | 85
percentage of total Hb | 93.2 [91.9 to 93.9] | 90.8 [85.7 to 93.7] | 58.0 [51.0 to 93.5] | 69.0 [47.3 to 93.5]
Statistical Analysis 1: Comparison: Only Cord-RBC vs Only adult_RBC vs Both Cord-RBC and adult_RBC; Group comparison is carried out among HbF values grouped according to the transfusion regimen (only cord blood transfusions, only adult transfusions, both cord and adult transfusions); Test type: Superiority; p < 0.0001, Kruskal-Wallis

2. Secondary Outcome: Post-transfusion Hematocrit (Htc) Change
Description: Change from baseline of Htc observed after either adult-RBC or cord-RBC transfusions. To this purpose, analysis was carried out between the two groups of RBC transfusions and patients were accordingly redistributed.
Time Frame: From enrollment to last HbF assessment occurring at 36 weeks, discharge or death
Population: Eight patients received 13 cord-RBC units and 9 patients received 18 adult-RBC units. Change of hematocrit value after each transfusion was recorded.
Measure: Median (Inter-Quartile Range); unit: percentage of total volume
Units Other Than Participants: number of transfusions
Groups:
- Cord-RBC Transfusions: top up transfusions obtained from cord blood of healthy full term neonates.
- Adult-RBC Transfusions: top up transfusions obtained from adult blood donors
Arm/Group | Cord-RBC Transfusions | Adult-RBC Transfusions
Number analyzed (Participants) | 8 | 9
Number analyzed (number of transfusions) | 13 | 18
percentage of total volume | 9.0 [6.5 to 12.0] | 11.5 [7.7 to 16]
Statistical Analysis 1: Comparison: Cord-RBC Transfusions vs Adult-RBC Transfusions; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.165

3. Secondary Outcome: Intervals Between Transfusions
Description: Number of days between two consecutive transfusions.To this purpose, analysis was carried out between the two groups of RBC transfusions and patients were accordingly redistributed.
Time Frame: From enrollment to the last HbF assessment occurring at 36 weeks, discharge or death
Population: Eight patients received a total number of 13 cord-RBC trasfusions and 9 patients received a total number of 18 adult -RBC transfusions. The intervals between two consecutive transfusions was recorded for each type of RBC unit.
Measure: Median (Inter-Quartile Range); unit: days
Units Other Than Participants: number of transfusions
Arm/Group | Cord-RBC Transfusions | Adult-RBC Transfusions
Number analyzed (Participants) | 8 | 9
Number analyzed (number of transfusions) | 13 | 18
days | 8.0 [5.0 to 18.5] | 7.0 [3.0 to 14.0]
Statistical Analysis 1: Comparison: Cord-RBC Transfusions vs Adult-RBC Transfusions; Test type: Superiority; p < 0.05, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 0.537

4. Secondary Outcome: Median Percentage of HbF at Last Assessment
Description: Median percentage of HbF at last HbF assessment. The last HbF measure was obtained at the completion of the 36 week of age, discharge or death.
Time Frame: From enrollment to the last HbF assessment occurring at 36 weeks, discharge or death
Population: Data recorded in all patient enetering the study were included in the analysis. Patients were grouped according to the type of RBC receved.
Measure: Median (Inter-Quartile Range); unit: % HbF
Units Other Than Participants: median HbF (%)
Arm/Group | Non Transfused | Cord-RBC Transfusions | Adult-RBC Transfusion | Cord- and Adult-RBC Transfusions
Number analyzed (Participants) | 13 | 3 | 4 | 5
Number analyzed (median HbF (%)) | 224 | 46 | 68 | 140
% HbF | 92.3 [91.0 to 93.4] | 90.6 [85.6 to 93.6] | 53.6 [48.8 to 92.7] | 62.0 [47.4 to 92.3]
Statistical Analysis 1: Comparison: Cord-RBC Transfusions vs Adult-RBC Transfusion vs Cord- and Adult-RBC Transfusions; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: From enrollment to postmenstrual age of 36 weeks.
Description: All cause mortality
Groups:
- Non-transfused: 13 preterm neonates non receiving transfusions
- Only Cord-TBC: 3 neonates receiving only cord-RBC
- Only Adult-RBC: 4 neonates receiving only adult-RBC
- Both Cord- and Adult-RBC: 5 neonates receiving both RBC types
Arm/Group | Non-transfused | Only Cord-TBC | Only Adult-RBC | Both Cord- and Adult-RBC
All-Cause Mortality (participants affected / at risk) | 0/13 | 1/3 | 1/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/13 | 3/3 | 3/4 | 5/5
Other Adverse Events (participants affected / at risk) | 0/13 | 0/3 | 0/4 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Non-transfused (N=13) | Only Cord-TBC (N=3) | Only Adult-RBC (N=4) | Both Cord- and Adult-RBC (N=5)
documented infections (Infections and infestations) | 0 | 1 | 1 | 3
Retinopathy stage II-III (Eye disorders) | 1 | 1 | 1 | 4
Necrotizing enterocolitis (Gastrointestinal disorders) | 0 | 1 | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/13/NCT03764813/Prot_SAP_ICF_000.pdf